CLINICAL TRIAL: NCT02392793
Title: A Phase I Study of Talazoparib (BMN 673) Plus Irinotecan With or Without Temozolomide in Children With Refractory or Recurrent Solid Malignancies
Brief Title: Talazoparib Plus Irinotecan With or Without Temozolomide in Children With Refractory or Recurrent Solid Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: St. Jude Children's Research Hospital (Other)
Collaborators: BioMarin Pharmaceutical (Industry); Alliance Pharma (Unknown); Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BMNIRN; NCI-2015-00255 (Registry Identifier: NCI Clinical Trial Registration Program)
Record Dates: First submitted 2015-03-06; First posted 2015-03-19 (Estimated); Last update posted 2021-02-09 (Actual); Status verified 2021-02

CONDITIONS: Childhood Solid Tumors
MeSH Terms: interventions — talazoparib; Irinotecan; Temozolomide; Filgrastim; Granulocyte Colony-Stimulating Factor; pegfilgrastim

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A: Talazoparib Plus Irinotecan (Active Comparator): Talazoparib will be administered orally on day 1 either once or twice per day depending on the dose level of the enrolled patient. Both oral talazoparib and IV irinotecan will then be administered daily, on days 2-6. Each cycle will last 21 days. Filgrastim or peg-filgrastim will be given following the last dose of chemotherapy.
  Arm A is closed to enrollment.
  Interventions: Drug: Talazoparib; Drug: Irinotecan; Drug: Filgrastim; Drug: Peg-filgrastim
- Arm B: Talazoparib Plus Irinotecan Plus Temozolomide (Active Comparator): Once the maximum tolerated doses (MTDs) for talazoparib and irinotecan are determined, a second arm of the study will open administering talazoparib, irinotecan and temozolomide. Talazoparib will be given orally, days 1-6. Intravenous irinotecan and oral temozolomide will be given days 2-6. Filgrastim or peg-filgrastim will be given following the last dose of chemotherapy.
  Interventions: Drug: Talazoparib; Drug: Irinotecan; Drug: Temozolomide; Drug: Filgrastim; Drug: Peg-filgrastim

INTERVENTIONS:
Drug: Talazoparib — Given orally once or twice on day 1 (depending on the dose level), then daily on days 2-6.
  Other Names: BMN 673
Drug: Irinotecan — Given intravenously daily, days 2-6 immediately following the talazoparib dose.
  Other Names: Camptosar®
Drug: Temozolomide — Given orally daily. Dose to be determined after MTD established with talazoparib plus irinotecan.
  Other Names: Temodar
  Arms: Arm B: Talazoparib Plus Irinotecan Plus Temozolomide
Drug: Filgrastim — Given subcutaneously (SubQ) once per day starting 24-36 hours after last dose of chemotherapy and continuing until post-nadir ANC is >2,000/μL, unless peg-filgrastim is given.
  Other Names: G-CSF; Neupogen®
Drug: Peg-filgrastim — Given subcutaneously (SubQ) once per day starting 24-36 hours after last dose of chemotherapy and continuing until post-nadir ANC is >2,000/μL, unless filgrastim is given.
  Other Names: Pegylated filgrastim; Neulasta®

SUMMARY:
The drug, talazoparib, seems to work against cancer in test tubes and animals by preventing DNA repair in damaged cells leading to their death. Investigators do not know if talazoparib combined with irinotecan will work in humans. Talazoparib has been used in only a small number of adults and children, and there is much not yet known about it.

In Arm A of this study, investigators seek to find the safest dose of irinotecan to give with talazoparib to children and young adults. In a phase I study, different dose levels of drug may be tested. The first 2 or 3 patients will be given a dose, and if none of them has a bad side-effect, the next 2 or 3 patients will be given a higher dose. No temozolomide will be given in in Arm A.

The experimental drug combination of talazoparib and irinotecan will be tested in the hopes of finding a treatment that may be effective against recurrent or refractory solid tumors. The goals of study Arm A are:

* To determine whether the combination of talazoparib and irinotecan is a beneficial treatment for your cancer;
* To learn what kind of side effects talazoparib can cause;
* To learn what kind of side effects talazoparib in combination with irinotecan can cause;
* To learn more about the biology of talazoparib in children diagnosed with solid tumors.

The purpose of Arm B is to to find the safest doses of irinotecan and temozolomide to give with talazoparib to children and young adults with a solid malignancy.. Talazoparib belongs to a family of drugs called "poly ADP ribose polymerase or PARP inhibitors." Irinotecan and temozolomide belong to a family of drugs called "DNA damaging agents."

There are two arms of this trial, A and B. In this study, investigators hope that irinotecan (administered in Arm A) and irinotecan plus temozolomide (administered in Arm B) will damage the DNA of the cancer cells. Then, talazoparib (which is a PARP inhibitor) will block the repair of the cancer cell's damaged DNA, causing the cancer cell to die (a process called "apoptosis").

There are different types of cancers found in children and young adults which appear to be vulnerable to the combination of chemotherapy agents that will be given in this study. Work carried out in the lab show that these agents may be very promising in the treatment of ewing sarcoma, germ cell tumors, wilms tumor, medulloblastoma and possibly neuroblastoma.

DETAILED DESCRIPTION:
In Arm A of this study, talazoparib will be administered orally on day 1 either once or twice per day depending on the dose level of the enrolled participant. Both oral talazoparib and intravenous (IV) irinotecan will then be administered daily, on days 2-6. Each cycle will last 21 days.

Once the maximum tolerated doses (MTDs) for talazoparib and irinotecan are determined, a second arm of the study (Arm B) will open administering talazoparib, irinotecan and temozolomide. Talazoparib will be given orally, on days 1-6. Intravenous irinotecan and oral temozolomide will be given on days 2-6. The study will estimate the maximum tolerated doses, describe the toxicities of therapy, estimate the response rate and characterize the pharmacokinetics of the combined talazoparib plus irinotecan with or without temozolomide.

This study is a traditional dose escalation study using a standard 3+3 phase I design. In Arm A, six or more dose levels will be evaluated for the combination of talazoparib and irinotecan. Once the MTDs of Arm A are determined, Arm B will open and evaluate the combination of talazoparib, irinotecan and temozolomide.

PRIMARY OBJECTIVES - ARM A

* To estimate the maximum tolerated doses (MTDs) of talazoparib (daily, days 1-6) combined with irinotecan (daily, days 2-6) given every 21 days in children with refractory or recurrent solid malignancies.
* To identify and describe the dose limiting toxicities of talazoparib and irinotecan administered in combination to patients with refractory or recurrent solid malignancies.

PRIMARY OBJECTIVES - ARM B

* To estimate the maximum tolerated dose (MTD) of temozolomide (given daily, days 2-6) when combined with talazoparib (daily, days 1-6) and irinotecan (daily, days 2-6) given every 21 days in children with refractory or recurrent solid malignancies.
* To identify and describe the dose limiting toxicities of temozolomide, talazoparib and irinotecan administered in combination to patients with refractory or recurrent solid malignancies.

SECONDARY OBJECTIVES

* To estimate the response rate, within the confines of a phase I study, to talazoparib plus irinotecan and talazoparib plus irinotecan and temozolomide administered in combination in pediatric patients with refractory or recurrent solid malignancies.
* To characterize the pharmacokinetics of talazoparib plus irinotecan and talazoparib plus irinotecan and temozolomide when given in combination to children with refractory or recurrent solid malignancies.

ELIGIBILITY:
INCLUSION CRITERIA:

* Patients with refractory or recurrent solid tumors for which there is no standard therapy are eligible. Patients must have had histologic verification of malignancy at original diagnosis or at the time of relapse.
* 12 months - 25 years at the time of enrollment on study.
* Patients must have a BSA of ≥ 0.42 m^2 at the time of study enrollment due to capsule strength(s).
* Patients must have either measureable or evaluable disease.
* Life expectancy must be at least 8 weeks.
* Performance status: Karnofsky ≥ 50 for patients > 16 years of age; Lansky ≥ 50 for patients ≤ 16 years of age.
* Prior therapy: Patients who have received prior therapy with an irinotecan-based or temozolomide-based regimen are eligible. Patients who have received prior therapy with a PARP inhibitor other than talazoparib are eligible; however, patients who have progressed on a PARP inhibitor plus irinotecan regimen are not eligible.
* Organ function: Must have adequate organ and bone marrow function as defined by the following parameters:

  * Patients with solid tumors not metastatic to bone marrow:
  * Peripheral absolute neutrophil count (ANC) ≥1,000/mm^3
  * Platelet count ≥ 100,000/mm^3 (no transfusion within 7 days of enrollment)
  * Hemoglobin ≥ 9 g/dL (with or without support)
  * Patients with solid tumors metastatic to bone marrow will be eligible for study but not evaluable for hematologic toxicity. These patients must not be known to be refractory to red cell or platelet transfusions. At least 2 of every cohort of 3 patients must be evaluable for hematologic toxicity. If dose limiting hematologic toxicity is observed at any dose level, all subsequent patients enrolled must be evaluable for hematologic toxicity.
  * Adequate renal function defined as: Serum creatinine concentration ≤3x the institutional upper limit of normal (ULN) or creatinine clearance or radioisotope GFR ≥ 70ml/min/1.73m^2.
  * Adequate liver function defined as: For Part A participants: normal liver function as defined by SGPT (ALT) concentration ≤5x the institutional ULN, a total bilirubin concentration ≤2x the institutional ULN for age, and serum albumin ≥ 2g/dL.
  * Adequate liver function defined as: For Part B participants: normal liver function as defined by SGPT (ALT) concentration < 2.5 times institutional ULN, a total bilirubin concentration ≤ 1.5 times the institutional ULN for age, and serum albumin ≥ 2 g/dL.
* Patients must have fully recovered from the acute toxic effects of chemotherapy, immunotherapy, surgery, or radiotherapy prior to entering this study:

  * Myelosuppressive chemotherapy: Patient has not received myelosuppressive chemotherapy within 3 weeks of enrollment onto this study (6 weeks if prior nitrosourea).
  * Hematopoietic growth factors: At least 7 days must have elapsed since the completion of therapy with a growth factor. At least 14 days must have elapsed after receiving pegfilgrastim.
  * Biologic (anti-neoplastic agent): At least 7 days must have elapsed since completion of therapy with a biologic agent. For agents that have known adverse events occurring beyond 7 days after administration, this period prior to enrollment must be extended beyond the time during which adverse events are known to occur.
  * Monoclonal antibodies: At least 3 half-lives must have elapsed since prior therapy that included a monoclonal antibody.
  * Radiotherapy: At least 2 weeks must have elapsed since any irradiation; at least 6 weeks must have elapsed since craniospinal RT or substantial bone marrow irradiation.
* All patients and/or their parents or legally authorized representatives must sign a written informed consent. Assent will be obtained, when appropriate, according to institutional guidelines.

EXCLUSION CRITERIA:

* Pregnant or breastfeeding.

  * If sexually active and with childbearing potential, must agree to use effective method of contraception, such as intrauterine device, bilateral tubal ligation for ≥ 6 months before randomization, partner vasectomized for ≥ 6 months before randomization, and sexual abstinence when in relation to the preferred and usual lifestyle of the subject.
  * Male subjects must use a condom when having sex with a pregnant woman and when having sex with a woman of childbearing potential from the time of the first dose of study drug through 105 days after the last dose of study drug.
  * Contraception should be considered for a nonpregnant female partner of childbearing potential.
  * Male subjects with partners of childbearing potential must use a condom and contraception should be considered for the female partner from the time of the first dose of study drug through 105 days after the last dose of study drug.
  * Male subjects whose partners are pregnant should use condoms for the duration of the pregnancy.
  * Male and female subjects must agree not to donate sperm or eggs, respectively, from the first dose of study drug through 105 days and 45 days after the last dose of study drug, respectively (hormonal contraception is not allowed) prior to study entry, during treatment, and for 45 days after last dose of study drug.
  * Females considered not of childbearing potential include those who are surgically sterile (bilateral salpingectomy, bilateral oophorectomy, or hysterectomy) or who are post menopausal, defined as: < 55 years of age with no spontaneous menses for ≥ 12 months before randomization and with a postmenopausal follicle stimulating hormone (FSH) concentration > 30 IU/L (or meeting criteria for post-menopausal status by the local laboratory).
  * If females with childbearing potential, a negative serum pregnancy test at Screening and willing to have additional serum and urine pregnancy tests during the study
  * Note: Females without childbearing potential include those in menopause ≥2 years, with tubal ligation ≥1 year before screening, or with total hysterectomy.
* Concomitant medications

  * Corticosteroids: Patients receiving corticosteroids that have not been on a stable or decreasing dose for at least 7 days prior to enrollment are not eligible.
  * Investigational drugs: Patients cannot receive other investigational drugs while on this study.
  * Anti-GVHD drugs post-transplant: Patients receiving cyclosporine, tacrolimus or other GVHD agents are not eligible.
* Prior treatment with talazoparib.
* Unable to swallow capsules.
* Active, uncontrolled infection.
* Prior solid organ transplant.
* Prior total body irradiation (TBI).
* Unwilling or unable to comply with the safety monitoring requirements of this protocol.

Ages: 12 Months to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 43 (Actual)
Dates: Start 2015-03-25 (Actual); Primary Completion 2019-02-20 (Actual); Study Completion 2019-08-30 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) of talazoparib combined with irinotecan | After first cycle (21 days) therapy of patients of Arm A.
  This study is a traditional dose escalation study using a standard 3+3 phase I design to define the MTD. Six or more dose levels will be evaluated for the combination of talazoparib and irinotecan. Each cycle will last 21 days with talazoparib given daily on days 1-6 and irinotecan given daily on days 2-6.
Dose-limiting toxicities (DLT) of talazoparib combined with irinotecan | After first cycle (21 days) therapy of patients of Arm A.
  Dose-limiting toxicities defined in the first cycle of the combination of talazoparib and irinotecan will be summarized for patients treated at each dose level with DLTs type and grade.
Maximum tolerated dose (MTD) of temozolomide combined with talazoparib | After first cycle (21 days) therapy of patients of Arm B.
  Once the MTD is defined for the combination of talazoparib plus irinotecan in Arm A, then temozolomide will be added to make a triple drug combination, talazoparib plus irinotecan and temozolomide. This is a traditional dose escalation study using a standard 3+3 phase I design to define the MTD. Six or more dose levels will be evaluated for the combination of talazoparib plus irinotecan and temozolomide. Each cycle will last 21 days with talazoparib given daily on days 1-6 and irinotecan and temozolomide given daily on days 2-6.
Dose-limited toxicities (DLT) of combination therapy with temozolomide, talazoparib and irinotecan | After first cycle (21 days) therapy of patients of Arm B.
  DLT defined in the first cycle of the combination of talazoparib plus irinotecan and temozolomide will be summarized for patients treated at each dose level with DLTs type and grade.

SECONDARY OUTCOMES:
Response rate | After 34 cycles of therapy (approximate 24 months).
  We will provide summary statistics for the best overall response (complete response, partial response, stable disease and progressive disease) of patients experienced during treatment.
Irinotecan Cmax | days 1 and 5 (week 1) of course 1
  A population average value and variance will be reported for week 1 of course 1
Talazoparib Cmax | days 1 and 5 (week 1) of course 1
  A population average value and variance will be reported for week 1 of course 1
Irinotecan AUC | days 1 and 5 (week 1) of course 1
  A population average value and variance will be reported for week 1 of course 1
Talazoparib AUC | days 1 and 5 (week 1) of course 1
  A population average value and variance will be reported for week 1 of course 1
Irinotecan Clearance | days 1 and 5 (week 1) of course 1
  A population average value and variance will be reported for week 1 of course 1
Talazoparib Clearance | days 1 and 5 (week 1) of course 1
  A population average value and variance will be reported for week 1 of course 1
Irinotecan Tmax | days 1 and 5 (week 1) of course 1
  A population average value and variance will be reported for week 1 of course 1
Talazoparib Tmax | days 1 and 5 (week 1) of course 1
  A population average value and variance will be reported for week 1 of course 1
Irinotecan t1/2 | days 1 and 5 (week 1) of course 1
  A population average value and variance will be reported for week 1 of course 1
Talazoparib t1/2 | days 1 and 5 (week 1) of course 1
  A population average value and variance will be reported for week 1 of course 1

CONTACTS AND LOCATIONS:
Overall Officials: Sara M. Federico, MD, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols